CLINICAL TRIAL: NCT01006200
Title: Factors to Obstructive Granulation Tissue Formation After Ultraflex Stenting in Benign Tracheal Narrowing
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Fu-Tsai Chung, Department of Thoracic Medicine, Chang Gung Memorial Hospital
Other Study IDs: 97-1411B
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: granulation tissue; benign; tracheal stenosis; ultraflex; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Structural /dynamic airway obstruction: Obstructive granulation tissue formation after SEMS implantation was defined as granulation tissue obstructing the lumen of the SEMS under bronchoscopic examination.

SUMMARY:
This study is aimed to determine factors leading to obstructive granulation tissue formation after placement of Self-Expandable Metallic Stent (SEMS) in patients with benign tracheal diseases.

DETAILED DESCRIPTION:
From August 2001 to September 2007, patients with benign tracheal stenosis who underwent endoscopic tracheal stent placements at the Chang Gung Memorial Hospital, a university-affiliated hospital in Northern Taiwan, were evaluated.

Definition of airway conditions Dynamic collapse (tracheao-malacia) was defined as tracheal lumen narrowing on expiration under bronchoscopic examination. Structural tracheal stenosis was defined as tracheal stenosis excluding dynamic collapse. Etiologies of structural tracheal stenosis were post-intubation or tracheostomy, post-tuberculosis infection, granulation tissue formation cause previous SEMS re-stenosis, previous SEMS fracture, corrosive injury with stricture, mediastinitis cause airway stricture, and goiter compression.

Obstructive granulation tissue formation after SEMS implantation was defined as granulation tissue obstructing the lumen of the SEMS under bronchoscopic examination, including the proximal and distal ends.

Significant variables, such as structural obstruction airway before SEMS implantation was entered into a forward logistical regression analysis to determine the net effect of each predictor while controlling the net effects of others to obstructive granulation tissue formation. Obstructive granulation tissue formation curves between patients with and those without structural tracheal stenosis before SEMS implantation were compared by log rank test.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* benign tracheal obstruction,
* receive Ultraflex metallic stent placement under flexible bronchoscopy.

Exclusion Criteria:

* malignant diseases,
* feasibility to receive surgical treatment or silicon stent placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign tracheal stenosis who underwent endoscopic tracheal stent placements at the Chang Gung Memorial Hospital, a university-affiliated hospital in Northern Taiwan, were evaluated.
  Chest surgeon were routinely consulted to evaluate feasibility of silicon stent placement in benign airway obstruction. All patients in our study were those unsuitable to receive silicon stent placement.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2001-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
factors to obstructive granulation tissue formation | time from stent placement to granualtion tissue formation after metallic stent placement in benign tracheal obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tsai Chung, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Madden BP, Stamenkovic SA, Mitchell P. Covered expandable tracheal stents in the management of benign tracheal granulation tissue formation. Ann Thorac Surg. 2000 Oct;70(4):1191-3. doi: 10.1016/s0003-4975(00)01555-1. PMID 11081868
- [Background] Lin SM, Lin TY, Chou CL, Chen HC, Liu CY, Wang CH, Lin HC, Yu CT, Lee KY, Kuo HP. Metallic stent and flexible bronchoscopy without fluoroscopy for acute respiratory failure. Eur Respir J. 2008 May;31(5):1019-23. doi: 10.1183/09031936.00099507. Epub 2008 Jan 9. PMID 18184680
- [Background] Kuo CH, Lin SM, Chen HC, Chou CL, Yu CT, Kuo HP. Diagnosis of peripheral lung cancer with three echoic features via endobronchial ultrasound. Chest. 2007 Sep;132(3):922-9. doi: 10.1378/chest.06-3106. Epub 2007 Jul 23. PMID 17646234